CLINICAL TRIAL: NCT03173898
Title: Periodontal Ligament Injection Versus Routine Local Infiltration, for the Non-surgical Single Posterior Maxillary Permanent Tooth Extraction: Comparative Double Blinded Randomized Clinical Study
Brief Title: PDL Anesthesia Versus Local Infiltration
Acronym: PDL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Mohammad H Al-Shayyab, Associate Professor, Assisstant Dean, Principal Investigator, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: RF: 10/2015/15791
Record Dates: First submitted 2017-05-28; First posted 2017-06-02 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Anesthesia, Local
Keywords: PDL Injection; Infiltration; Anesthesia; Extraction

STUDY DESIGN:
Intervention Model Description: a prospective randomized double blinded, split mouth study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The method of anesthesia used for the left or right sides was blinded to the patient and determined randomly by the same surgeon (MA) who was not involved in the extraction. the extraction procedure was randomly commenced by the same resident who was blinded to the anesthetic technique administered randomly by the surgeon.participiants were also blinded to the type of technique applied on each side.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- primary periodontal ligament anesthesia (Experimental): PDL anesthesia versus local infiltration
  Interventions: Procedure: PDL anesthesia versus local infiltration
- local infiltration (Active Comparator): PDL anesthesia versus local infiltration
  Interventions: Procedure: PDL anesthesia versus local infiltration

INTERVENTIONS:
Procedure: PDL anesthesia versus local infiltration — Every patient received the recommended volumes of 2% lidocaine with 1:100.000 epinephrine for PDL injection on the experimental side, and for local infiltration on the control side. A Visual Analogue Scale (VAS) was used to describe the pain felt during injection.

SUMMARY:
The literature concerning the success and pain scores of PDL injection technique compared with other techniques remains controversial; whereas some studies found no significant difference in pain scores between local infiltration and PDL injection, other older studies found that pain during administration of PDL injection was described by the majority of patients either as greater than local infiltration6, or as negligible or as a less painful injection compared with other injection techniques. The aim of this study was to evaluate the efficacy of and patients' subjective responses to the PDL injection technique as compared to the traditional infiltration injection, for the non-surgical extraction of one posterior maxillary permanent tooth.

DETAILED DESCRIPTION:
Aim: The aim of this study was to evaluate the efficacy of and patients' subjective responses to the periodontal ligament (PDL) anesthetic injection as compared to the traditional infiltration injection, for the non-surgical extraction of one posterior maxillary permanent tooth. Methods: All patients scheduled for non-surgical symmetrical maxillary posterior permanent teeth extraction in the Department of Oral and Maxillofacial Surgery (OMFS) at the University of Jordan Hospital, Amman, Jordan, over a-seven-month period, were invited to participate in this prospective randomized double blinded, split mouth study. Every patient received the recommended volumes of 2% lidocaine with 1:100.000 epinephrine for PDL injection on the experimental side, and for local infiltration on the control side. A Visual Analogue Scale (VAS) and a Verbal Rating Scale (VRS) were used to describe the pain felt during injection and extraction, respectively. Statistical significance was based on probability values of <0.05 and measured using Chi-Square and Student-t tests, and Nonparametric Mann-Whitney and Kruskal-Wallis tests.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria were: patients who were fit for surgery under LA (classified by the American Society of Anaesthesiologists (ASA) as ASA I-ASA III); patients exhibiting full understanding of given oral instructions; and bilateral symmetrical posterior maxillary permanent teeth referred for non-surgical extractions under LA.

Exclusion Criteria:

Exclusion criteria were: the presence of acute dento-alveoalr infection; patients requiring conscious sedation or general anesthesia; patients unwilling to participate in the study; patients with ASA greater than III; patients on anti-inflammatory or recreational drugs; and patients requiring more than two additional injections in one or both sides for incomplete anesthesia.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-07-06 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
the Visual Analogue Scale (VAS) scores for injections pain | 5 minutes
  The VAS composed of a 100-mm line and allowed the patient to score the pain experienced during injections as low moderate and high

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad H Al-Shayyab, Fellowship, Principal Investigator — The University of Jordan

IPD SHARING:
Plan to Share IPD: Undecided